CLINICAL TRIAL: NCT04862026
Title: The Influence of Telemonitoring on the Development of Clinical Events and Improving the Quality of Life of Patients With Acute Coronary Syndrome (TeleCor)
Brief Title: Telemonitoring of Patients With Acute Coronary Syndrome
Acronym: TeleCor
Status: Suspended | Type: Observational
Why Stopped: Technical difficulties of the developer
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1
Record Dates: First submitted 2021-04-14; First posted 2021-04-27 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome, telemonitoring
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telemonitoring group: The telemonitoring group will be connected to electronic medical systems, through which medical workers will remotely assess clinical and emotional status, adherence to drug therapy, and carry out nutritional adjustments.
- Control group: Patients with standard administration.

SUMMARY:
It is planned to enroll 950 patients in an open, prospective, randomized study to assess the impact of telemonitoring on the development of clinical events and improve the quality of life of patients with acute coronary syndrome. The duration of the study is 365 days, of which 180 days are enrollment of patients, 180 days are observation. The study of patients will include the collection of anamnesis, assessment of the clinical status of patients using special questionnaires, data of objective, laboratory and instrumental examinations. The instrumental complex of the examination will include: electrocardiography (ECG), 6-minute walk test (6MWT), Holter ECG monitoring (HMECG), echocardiography, veloergometry (VEM), assessment of the actual nutrition Nutrilogic, autogeneration of an individual diet (Nutrilogic), weekly telemonitoring. Laboratory examination includes: biochemical blood test. The main objectives of the study are to study the effect of telemonitoring on mortality from cardiovascular diseases (CVD), as well as the number of readmissions for cardiovascular pathology in patients with ACS. The secondary endpoints of the study include quality of life as measured by the HeartQol questionnaire and adherence to ambulatory monitoring.

DETAILED DESCRIPTION:
Purpose of the study: to study the effect of telemonitoring on the development of clinical events and improving the quality of life of patients with ACS.

Research objectives:

1. Improving the effectiveness of medical care in patients who have undergone ACS: increasing the level of compliance of patients, increasing the level of medical awareness of patients, reducing the number of unmotivated requests for medical care, reducing the time to achieve the observed targets, reducing the proportion of complications, reducing the number of destabilizing conditions with further inpatient treatment, optimization of the workload on medical personnel.
2. Creation of a unified methodology for remote observation using telemedicine technologies in patients with ACS.
3. Creation of a unified model of remote nutrition correction in patients after ACS.

Number of volunteers: statistically equivalent groups by sex and age, 950 subjects (475 per group). The number of volunteers who completed the study was 712 subjects (75% of the total number of patients).

365 days: 6 months enrollment, 6 months follow-up.

Inclusion criteria:

* Signed informed consent;
* Age 18 - 80 years old.
* Diagnosis:

  * Acute myocardial infarction (I21.0, I21.1, I21.2, I21.3, I21.4, I21.9)
  * Unstable angina (I20.0) Recurrent myocardial infarction (I22.0, I22.1, I22.8, I22.9)

Exclusion criteria:

* Lack of technical equipment to connect to remote monitoring programs;
* Severe cognitive dysfunction - dementia leading to maladjustment in everyday life;
* Mental illness in the acute stage;
* Oncological diseases requiring radiation and chemotherapy during the period of this study, as well as the corresponding stages of T3-4N2-3M1;
* Lack of technical ability to take part in telemonitoring (do not have the skills to work on a smartphone, computer, tablet, there is no appropriate technical means);
* Participation in other clinical studies to assess the effectiveness of pharmacological drugs.

Exclusion criteria:

* Infection with SARS-CoV-2 with laboratory confirmation during the period of this study;
* Acute coronary syndrome that developed in the hospital after surgery / intervention;
* The emergence during the observation of the need for surgical (not counting myocardial revascularization) or chemotherapy treatment;
* Severe injuries (including craniocerebral), impeding observation according to the study protocol.

Primary endpoint (combined):

1. a) Death from cardiovascular causes and / or b) Repeated hospitalizations for SS pathology
2. The number of episodes requiring emergency or urgent care without hospitalization (calls to the emergency room for complaints from the cardiovascular system)

Secondary endpoints:

1. Quality of life according to the HeartQol questionnaire.
2. Commitment to outpatient monitoring - is determined by the number of participants who voluntarily left the study, by the percentage of results obtained - surveys in electronic form.
3. Tolerance to physical activity (any increase in walking distance according to 6MWT, VEM according to indications).

Any decrease in body weight (weight, BMI) any decrease in waist circumference. The study of patients will include the collection of anamnesis, assessment of the clinical status of patients using special questionnaires, data of objective, laboratory and instrumental examinations. The instrumental complex of the examination will include: electrocardiography (ECG), 6-minute walk test (6MWT), Holter ECG monitoring (HMECG), echocardiography, veloergometry (VEM), assessment of the actual nutrition Nutrilogic, autogeneration of an individual diet (Nutrilogic), weekly telemonitoring. Laboratory examination includes: biochemical blood test.

Randomization by means of envelopes.

It is planned to create in advance a database of identification numbers (hereinafter - ID) in the amount corresponding to the planned set of patients (950 ID). Further, these numbers will be divided into two groups with an equal number of IDs in each:

* Outpatient observation with connection to the telemonitoring program - 475 ID
* Outpatient monitoring without connecting to the telemonitoring program - 475 ID Each ID number will be placed in an individual envelope and sealed. In accordance with the agreement on the number of patients to be included in the study, each specific healthcare facility will be provided with sealed envelopes in the required volume, taking into account the equal distribution of volunteers into 2 groups. After opening the envelope, the patient is assigned this ID, and the patient is assigned to the corresponding ID group.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age 18 - 80 years old.
* Diagnosis:

  * Acute myocardial infarction (I21.0, I21.1, I21.2, I21.3, I21.4, I21.9)
  * Unstable angina (I20.0) Recurrent myocardial infarction (I22.0, I22.1, I22.8, I22.9)

Exclusion Criteria:

* Lack of technical equipment to connect to remote monitoring programs;
* Severe cognitive dysfunction - dementia leading to maladjustment in everyday life;
* Mental illness in the acute stage;
* Oncological diseases requiring radiation and chemotherapy during the period of this study, as well as the corresponding stages of T3-4N2-3M1;
* Lack of technical ability to take part in telemonitoring (do not have the skills to work on a smartphone, computer, tablet, there is no appropriate technical means);
* Participation in other clinical studies to assess the effectiveness of pharmacological drugs;
* Infection with SARS-CoV-2 with laboratory confirmation during the period of this study;
* Acute coronary syndrome that developed in the hospital after surgery / intervention;
* The emergence during observation of the need for surgical (not counting myocardial revascularization) or chemotherapy treatment;
* Severe trauma (including craniocerebral) impeding observation according to the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome who have undergone the hospital stage of treatment are included in the study at the time of discharge. And then, at the outpatient stage after randomization, the first group receives standard assistance together with telemonitoring support, the second group - standard offline medical assistance.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Death or rehospitalizations Primary endpoint A | Upon completion, up to 6 months
  Death from cardiovascular causes and / or rehospitalizations for cardiovascular pathology
Emergency or urgent care without hospitalization | Upon completion, up to 6 months
  The number of episodes requiring emergency or urgent care without hospitalization (calls to the ambulance for complaints from the cardiovascular system)

SECONDARY OUTCOMES:
Quality of life according to the HeartQol questionnaire. | Upon completion, up to 6 months
  Health-related quality of life, symptoms, and functional status make up patient-reported outcomes
Commitment to outpatient monitoring | Upon completion, up to 6 months
  Commitment to outpatient monitoring - is determined by the number of participants who voluntarily left the study, by the percentage of results obtained - surveys in electronic form.
Tolerance to physical activity | Upon completion, up to 6 months
  Tolerance to physical activity (any increase in walking distance according to 6MWT, VEM according to indications).
Decrease in body weight | Upon completion, up to 6 months
  Any decrease in body weight (weight, BMI) any decrease in waist circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Morozov, Study Director — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Locations (1):
- City Clinical Hospital No. 13 of the Moscow City Health Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No